CLINICAL TRIAL: NCT01898065
Title: Evaluation of Hypoxia by PET With 18-FluoroMisonidazole During Radiation Therapy of Prostate Cancer
Brief Title: Evaluation of Hypoxia by PET With F-Miso in Radiation Therapy of Prostate Cancer
Acronym: HYPOXProstat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Poitiers University Hospital (Other); IASON Gmbh, Feldkirchner strasse 4, 8054 Graz-Seiesberg AUSTRIA (Unknown); Cyclopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC11-080; 2011-004582-32 (EudraCT Number)
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Adenocarcinoma
Keywords: Hypoxia; radiotherapy; PET with 18-F-MISO; MRI
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET imaging, 18 F-miso (Experimental): Single Arm study
  Interventions: Drug: 18-F-MISO

INTERVENTIONS:
Drug: 18-F-MISO — PET scan with the 18 Fluoro Misonidazole
  Other Names: 18 Fluoro Misonidazole

SUMMARY:
With functional imaging development, it becomes possible to increase radiation dose to radioresistant areas (located inside tumor volume) using radiotherapy dose-painting. This strategy is particularly suitable for prostate cancer where tumor hypoxia plays a major role in the resistance of these tumors to radiation.

In order to develop intratumoral hypoxia targeting by radiotherapy dose-painting areas, we should characterize changes in hypoxia before treatment and during radiotherapy.

* If hypoxia does not change during radiotherapy, radiotherapy dose-painting strategy by an "integrated" boost is performed.
* If hypoxia varied (increasing or incomplete regression), a "final" boost strategy of radiotherapy dose-painting(IMRT, stereotactic brachytherapy or high dose rate) after a first fractionated IMRT could be considered.

This study should show that PET imaging with fluoromisonidazole (18F-MISO) is an available tool to physicians in assessing tumor hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven prostate adenocarcinoma
* Absence of metastases (lymph node or bone)
* One or more tumor nodules seen on MRI and PET Choline.
* Intermediate Risk : Gleason 7 and PSA (prostate specific antigen)<20 ng / ml, T <T2c or Gleason 6 and PSA 10-20 ng / ml, T <T2c
* No concomitant hormonal treatment. (NB: the introduction of hormone therapy during radiotherapy before the second 18F-MISO is a criterion to study exit)
* Indication of radiotherapy up to a total dose> 70 Gy and 2 Gy/day fractions
* Signed Informed consent
* Social Insurance

Exclusion Criteria:

* Age < 18 years old
* Patient protected by law

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To characterize changes in tumor hypoxia (PET with 18F-MISO) during radiation therapy of prostate cancer. | 3 to 4 weeks after beginning of radiation therapy
  First PET-scan with 18-F-Miso done before radiation Second PET-scan with 18-F-Miso done 3 to 4 weeks after the beginning of radiation therapy.

SECONDARY OUTCOMES:
To compare hypoxia imaging (PET with 18F-MISO) with anatomical imaging (PET with 18F-choline) to study the feasibility of a tailored treatment. | before and 3 to 4 weeks after the begining of radiation therapy
  Images obtained with PET Choline and MRI (anatomical location) will be merge with images obtained by 18F-MISO PET to search hypoxia on these anatomical areas.

CONTACTS AND LOCATIONS:
Overall Officials: SUPIOT Stéphane, MD, Principal Investigator — ICO René Gauducheau
Locations (2):
- France (2):
  - CHU Poitiers, Poitiers
  - ICO Rene Gauducheau, Saint-Herblain

REFERENCES:
- [Result] Rasey JS, Koh WJ, Evans ML, Peterson LM, Lewellen TK, Graham MM, Krohn KA. Quantifying regional hypoxia in human tumors with positron emission tomography of [18F]fluoromisonidazole: a pretherapy study of 37 patients. Int J Radiat Oncol Biol Phys. 1996 Sep 1;36(2):417-28. doi: 10.1016/s0360-3016(96)00325-2. PMID 8892467
- [Result] Bentzen SM. Theragnostic imaging for radiation oncology: dose-painting by numbers. Lancet Oncol. 2005 Feb;6(2):112-7. doi: 10.1016/S1470-2045(05)01737-7. PMID 15683820
- See also: Sponsor web site — http://www.centregauducheau.fr/